CLINICAL TRIAL: NCT04409912
Title: SIroliMus Coated angioPlasty Versus Plain Balloon Angioplasty in the tREatment of dialySis acceSs dysfunctION (IMPRESSION)
Brief Title: Sirolimus Coated Angioplasty Versus Plain Balloon Angioplasty
Acronym: IMPRESSION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: National University Hospital, Singapore (Other); Sengkang General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/2896
Record Dates: First submitted 2020-04-24; First posted 2020-06-01 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: End Stage Renal Failure on Dialysis; Arteriovenous Graft Occlusion

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in a 1:1 ratio into either the treatment (SCB) arm or control (PB) arm. As above-elbow AVFs generally have larger vessel size and better outcomes compared to below-elbow AVFs, randomisation will be stratified by location of AVF (above vs below elbow) to ensure a more even distribution of AVF by location between both groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Dialysis centre staff and procedurist performing the intervention will also be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus coated balloon (Experimental): The trial product is MagicTouch sirolimus drug coated balloon (Concept Medical). Sirolimus will be transferred from the balloon to the vessel wall by inflating the sirolimus coated balloons at 2 minutes at rated burst pressure (typically 12 to 14ATM). All the lesions within the dialysis circuit with sirolimus coated balloon.
  Interventions: Device: Sirolimus coated balloon
- Plain balloon (Placebo Comparator): The plain balloon or placebo will not be coated. The plain balloon will be inflated at 2 minutes at rated burst pressure (typically 12 to 14 ATM). Plain balloon will be applied to all the narrowed segment of the dialysis circuit
  Interventions: Device: Plain balloon

INTERVENTIONS:
Device: Sirolimus coated balloon — Sirolimus has a high transfer rate to the vessel wall and effectively inhibit neointimal hyperplasia in the porcine coronary model. In coronary artery interventions, preliminary clinical studies using sirolimus coated balloon have shown excellent procedural and 6 month patency. The effectiveness of sirolimus coated balloon in patients with dialysis access dysfunction has been shown in a small pilot study in the salvage of thrombosed arteriovenous graft.
  When compared to Paclitaxel, sirolimus is cytostatic in its mode of action with a high margin of safety.
  Arms: Sirolimus coated balloon
Device: Plain balloon — Plain balloon angioplasty is the current standard therapy to treat stenosis in dialysis access. However, the mid and long term patency of plain balloon angioplasty in patients with end stage renal disease is poor. The average primary patency is around 40 to 50 percent at 1 year and multiple repeated angioplasty is required to maintain the patency of the vascular access.
  Arms: Plain balloon

SUMMARY:
A functioning dialysis access is critical to the delivery of hemodialysis therapy in patients with End Stage Renal Disease. Stenosis secondary to neo-intimal hyperplasia frequently occur within the dialysis access, resulting in dysfunction. Conventional balloon angioplasty is the current standard of care for treatment of stenosis but is associated with high rate of recurrence. Paclitaxel coated balloon has been shown to be superior to conventional balloon angioplasty in dialysis access interventions but recent meta-analysis has shown an increase in mortality when paclitaxel coated balloon and stents are used in lower limb angioplasty. Sirolimus coated angioplasty balloon are second generation drug coated balloon that have been shown to be effective in coronary artery interventions. Sirolimus is cytostatic in nature with good safety profile. In our pilot study, sirolimus coated balloon has been shown to be safe and effective in the salvaged of thrombosed arteriovenous graft. Therefore, the investigators are conducting a double-blinded, multi-center randomised control trial to compare the 6 month patency of arteriovenous fistula after intervention with sirolimus coated balloon versus conventional balloon angioplasty.

The investigators hypothesise that the addition of SCB after successful balloon angioplasty with conventional plain balloon is superior to conventional plain balloon angioplasty alone with decreased restenosis of the treated lesion, improved access circuit and treated lesion patency, and decreased number of interventions needed to maintain patency.

DETAILED DESCRIPTION:
Dialysis vascular accesses such as Arteriovenous Fistula (AVF) and Arteriovenous Grafts (AVG) are surgically created vasculatures used for hemodialysis in patients with End-Stage Renal Disease (ESRD). A functioning dialysis vascular access is critical to the delivery of life-saving hemodialysis (HD) treatment to these patients. Unfortunately, neointimal hyperplasia frequently occurs within the dialysis vascular access, resulting in stenosis, poor flow and thrombosis with loss of function. The durability of both AVF and AVG are poor, with an almost 50% failure rate after a median lifetime of 3 to 7 years for AVF and 12 to 18 months for AVG. Vascular access failure is the most common reason for hospitalization among HD patients. The global healthcare costs for treating vascular access-related complications amount to USD 18 billion, and in USD 1 billion in the US alone. These figures are set to increase, due to the increase in the prevalence of access interventions and hemodialysis patients globally. Singapore has one of the highest ESRD rates in the world and the investigators are facing an increasing number of patients with ESRD and the majority of the patients opting for hemodialysis as their treatment modality. As such, vascular access-related complication is set to be a major contribution of healthcare cost in our nation.

The current gold standard therapy for the treatment of stenosis in dialysis access is plain balloon angioplasty (BA). Despite its widespread availability and minimally invasive nature, the mid- and long-term patency with BA in patients with ESRD is poor. The reported average primary patency after BA is around 40-50% at 1 year. Multiple repeated angioplasty is required to maintain the patency of the vascular access. Hence, there is an urgent clinical need to improve the patency of dialysis vascular access.

Recently, the use of stents, in particular stent graft, has been shown to be superior to angioplasty for stenosis occurring at the site of venous anastomoses of an AVG. The incidence of patency of the treatment area was significantly greater in the stent-graft group than in the balloon-angioplasty group (51% vs. 23%, P<0.001), as was the incidence of patency of the access circuit (38% vs. 20%, P=0.008) at 6 months. For cephalic arch stenosis in AVF, the use of stent graft has also been shown to be superior to bare metal stent. The 6 month primary patency for stent graft and bare stent was 81.8 and 39.1%, respectively. One-year primary patency for stent graft and bare stent was 31.8 and 0.00%, respectively (P = 0.002). However, the use of stent graft for the management of dialysis vascular access is not without any concern. In particular, re-stenosis can occur within the stented segment (post stent 12-month primary patency is 46%), resulting in the need for repeat angioplasty. Future stent deployment in the re-stenotic segment may also not be feasible due to the presence of the stent. Moreover, the presence of a stent can impede future surgical revision or new access creation within the same vessel.

Paclitaxel-coated balloon angioplasty (PCBA) has also been shown recently to be superior to plain BA in the treatment of stenosis in dialysis vascular access. This is because the very intervention used to treat the underlying stenosis by plain BA can induce vascular injury and accelerate intimal hyperplasia, resulting in rapid restenosis and the need for repeated procedures to maintain vessel patency. By releasing Paclitaxel, which is an anti-proliferative drug, locally into the vessel wall during balloon contact, it will blunt the acceleration of intimal hyperplasia response, resulting in improved primary patency after angioplasty. Additionally, unlike stents, PCBA does not leave a permanent structure that may impede future surgical revision. In a small 40 patient pilot study, the primary unassisted patency in the PCBA group was significantly better than the plain BA group at 6 (70 % versus 25 %) and 12 months (35 % versus 5 %, p <0.001) respectively. Recent randomized control trials have also shown the superiority of PCBA over plain balloon angioplasty in the treatment of stenosis in dialysis vascular access. However, concerns had also arisen recently in the use of PCBA. In large lower limb studies involving the use of PCBA, meta-analysis had revealed an increased risk of death in patients that are treated with PCBA or paclitaxel-coated stent. This had led to warning from the United States Food and Drug Administration (FDA) and the issue of guidelines from the interventional societies

Sirolimus coated balloon (SCB) is the new generation of drug-eluting balloons available in the market. Compared to Paclitaxel, sirolimus is cytostatic in its mode of action with a high margin of safety. It has a high transfer rate to the vessel wall and effectively inhibits neointimal hyperplasia in the porcine coronary model. In the coronary artery interventions, preliminary clinical studies using SCB have also shown excellent procedural and 6-month patency.

The effectiveness of SCB in patients with dialysis access dysfunction has been shown in a small pilot study in the salvage of thrombosed AVG and investigators postulate that SCB will be a viable option in patients who requires treatment with drug-coated balloon.

The investigators aim to conduct a multicenter double-blinded randomized controlled trial to compare the 6 month unassisted patency rate of SCB angioplasty versus plain balloon angioplasty in the management of stenosis in arteriovenous fistula.

RECRUITMENT:

Patients with matured AVF (in use for more than 1 month) that are dysfunctional and are already scheduled to undergo balloon angioplasty will be considered for the trial. Patients will be consented if they fulfill the preliminary eligibility criteria and are agreeable to participate in the study. Once all the eligibility criteria are fulfilled, including angiographic criteria assessed on the day of the procedure, the patient is entered into the trial and randomised. Patients who are unsuitable for the trial will be treated in the conventional way with PB and considered as screen failure.

STUDY PROCEDURE:

The AVF will be assessed with ultrasound for possible access sites. All patients will undergo a fistulogram which is obtained by injection of contrast. The access site will be left to the discretion of the procedurist. The fistulogram should include the entire dialysis circuit from the arteriovenous anastomosis to the central veins. The suggested approach would include a fistulogram via an 18 Gauge cannula inserted into the arterialised vein. When there is no spontaneous reflux of contrast into the artery, reflux opacification of the arteriovenous (AV) anastomosis is achieved by injecting contrast during inflation of a blood pressure cuff or a tourniquet around the arm. Alternatively, a trans-radial or arterial approach may be used to obtain the fistulogram

Based on fistulogram findings, the access site will be placed up to the discretion of the procedurist. If an 18G cannula is used, it may be exchanged for a vascular sheath that is sized appropriately based on the planned balloon sizes). Alternatively, the 18G cannula may be removed and a new access site for intervention may be chosen. A new puncture will be performed with the insertion of a vascular sheath (sized appropriately according to planned balloon sizes). Two access sites (both antegrade and retrograde) may be needed in certain cases. A trans-radial or arterial approach may also be considered if necessary

In the event that opacification of the anastomosis was not earlier achieved even with inflation of a blood pressure cuff around the arm, it will be performed via contrast injection through a catheter in the feeding artery.

When there is more than 1 stenosis, all the lesions will be labelled and treated with conventional balloon angioplasty (from the AV anastomosis up to, but not including, the subclavian vein). Lesions are considered separate if they are separated by a gap of at least 2 cm. The lesion or lesions will be dilated with standard angioplasty that is sized similar to the adjacent reference vessel. Inflation time will be at least 1 minute per inflation. The balloon will be inflated to an appropriate inflation pressure as per institution standardised practice to achieve <30% residual stenosis and satisfactory thrill. If there is significant residual stenosis after angioplasty (defined as > 30% stenosis), repeat angioplasty with the same standard angioplasty balloon or a larger standard angioplasty balloon may be used at operator's discretion. High-pressure angioplasty balloon or cutting balloon may also be used, if necessary, in the event of resistant stenosis. In stenotic segment adjacent to aneurysmal segment, where the percentage of stenosis is difficult to determine, the treated segment should reach at least reach 6mm.

Randomisation occurs when all the lesions are treated adequately, defined as less than 30% residual stenosis after standard treatment.

Patients will be randomised to receive either the sirolimus coated balloon or plain balloon. Repeated angioplasty of the stenotic segments that were successfully treated (defined as less than 30% residual stenosis) will be performed using sirolimus coated balloon (for patient randomised into the sirolimus balloon arm) or plain/placebo balloon (for patients randomised into the placebo arm)

POST-PROCEDURE ULTRASOUND SCAN:

All participants will receive an ultrasound scan of their AVF after their procedure before discharge. The diameter of the vessel at the treated sites will be measured and documented. Brachial artery flow and flow within the outflow vein will also be measured and documented

* Patency definitions are defined based on SIR reporting standards (Gray et al., 2003):

Post-intervention target lesion patency:

Interval after intervention until the next re-intervention at or adjacent to the original treatment site or until the access is abandoned. Percutaneous or surgical treatments of a new arterial or venous outflow stenosis/occlusion (including access thrombosis) that do not involve or exclude the original lesion from the access circuit are compatible with lesion patency. The creation of new access that incorporates the target lesion into the new access circuit is also compatible with target lesion patency.

Post-intervention access circuit primary patency:

Interval following intervention until the next access thrombosis or repeated intervention. It ends with the treatment of a lesion anywhere within the access circuit, from the arterial inflow to the superior vena cava-right atrial junction.

Post-intervention access circuit assisted primary patency:

Interval after intervention until access thrombosis or surgical intervention that excludes the treated lesion from the access circuit. Percutaneous treatments of either restenosis/occlusion of the previously treated lesion or a new arterial or venous outflow stenosis/occlusion (excluding access thrombosis) are compatible with assisted primary patency.

Post-intervention access circuit secondary patency:

Interval after intervention until the access is surgically declotted, revised or abandoned. Thrombolysis and percutaneous thrombectomy are compatible with secondary patency.

^Complications will be categorised according to SIR definitions of minor or major complications (Aruny et al., 2003):

A major complication is defined as one that:

1. require therapy, minor hospitalisation (< 48 hours),
2. require major therapy, unplanned increase in the level of care, prolonged hospitalisation (>48 hours),
3. leads to permanent adverse sequelae, or
4. death

A minor complication is one that:

1. requires no therapy with no consequence,
2. requires nominal therapy with no consequence; includes overnight admission for observation only.

POST-PROCEDURE FOLLOW-UP ULTRASOUND SCAN OF AVF:

Patients will be followed-up at:

3 months (± 1 weeks): assessment of primary outcome 6 months (± 4 weeks): assess the target lesion and access circuit. 12 months (± 4 weeks): assess AVF patency and study closure

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 to 85 years
2. Patient who requires balloon angioplasty for dysfunction arteriovenous fistula
3. Matured AVF, defined as being in use for at least 1 month prior to angioplasty
4. 4. Successful angioplasty of the underlying stenosis, defined as less than 30% residual stenosis on Digital Subtraction Angiography (DSA) based on visual assessment of the operator and restoration of thrill in the AVF on clinical examination. (For concurrent asymptomatic or angiographically not significant central vein stenosis, patients can be included if no treatment is required.)

Exclusion Criteria:

1. Patient unable to provide informed consent
2. Thrombosed or partially thrombosed AVF
3. Presence of symptomatic or angiographically significant central vein stenosis who require treatment, with more than 30% residual stenosis post angioplasty
4. Patients who had underwent stent placement within the AVF circuit
5. Patient who are currently enrolled in other drug eluting balloon trials
6. Sepsis or active infection
7. Recent intracranial bleed or gastrointestinal bleed within the past 12 months
8. Allergy to iodinated contrast media, anti-platelet drugs, heparin or sirolimus
9. Pregnancy

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Primary patency of the AVF at 6 months | 6 months
  This is measured by the percentage of patients whose AVF remain patent at 6 months after the procedure

SECONDARY OUTCOMES:
Time taken to the next intervention | Through study completion, an average of 1 year
  The number of months from procedure to the next interventions. This will be track until study completion.
Treated lesion percent stenosis at 6 and 12 month ultrasound | 6 and 12 months
  Defined as percent stenosis relative to adjacent reference vessel, [1 - (minimum lesion diameter / reference vessel diameter)] x 100)
Treated lesion re-stenosis rate at 6 months | 6 months
  Defined as incidence of stenosis > 50% diameter of adjacent reference vessel segment
Number of repeat interventions to treated lesion at 6 and 12 months | 6 and 12 months
  How many repeat interventions to treated lesion at 6 and 12 months
Number of repeat interventions to maintain access circuit (including interventions to treated lesion) at 6 and 12 months | 6 and 12 months
  How many repeat interventions to maintain access circuit (including interventions to treated lesion) at 6 and 12 months
Treated lesion revascularisation free interval | anytime within 12 months study participation
  Defined as the interval from intervention to repeat clinically driven target lesion intervention
De nova stenosis detected on ultrasound scan at 3, 6 and 12 months | 3, 6 and 12 months
  Presence of De nova stenosis detected on ultrasound scan at 3, 6 and 12 months
Post intervention treated lesion patency at 3, 6 and 12 months | 3, 6 and 12 months
  Percentage of patients whose treated stenosis remains patent at 3, 6, and 12 months after the procedure. This is determined by the use of ultrasound imaging or angiogram or clinical examination.
Post-intervention primary patency at 3, 6 and 12 months | 3, 6 and 12 months
  Percentage of patients whose AVF remains patent and does not require any further interventions at 3, 6, and 12 months after the procedure. This is determined by the use of ultrasound imaging or angiogram or clinical examination.
Post-intervention assisted primary patency at 3, 6 and 12 months | 3, 6 and 12 months
  Percentage of patients whose AVF requires additional interventions to remains patent at 3, 6, and 12 months after the procedure. This is determined by clinical history during the study period
Post-intervention secondary patency at 3, 6 and 12 months | 3, 6 and 12 months
  Percentage of patients whose AVF has thrombosed and required additional procedure to restore flow at 3, 6, and 12 months after the procedure. This is determined by clinical history during the study period.
Complication rates at 1, 3, 6 and 12 months | 1, 3 6 and 12 months
  Complication rates at 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chieh Suai Tan, MD, Principal Investigator — Singapore General Hospital
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Sengkang General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roy-Chaudhury P, Sukhatme VP, Cheung AK. Hemodialysis vascular access dysfunction: a cellular and molecular viewpoint. J Am Soc Nephrol. 2006 Apr;17(4):1112-27. doi: 10.1681/ASN.2005050615. PMID 16565259
- [Background] Lee T, Roy-Chaudhury P. Advances and new frontiers in the pathophysiology of venous neointimal hyperplasia and dialysis access stenosis. Adv Chronic Kidney Dis. 2009 Sep;16(5):329-38. doi: 10.1053/j.ackd.2009.06.009. PMID 19695501
- [Background] Pantelias K, Grapsa E. Vascular access today. World J Nephrol. 2012 Jun 6;1(3):69-78. doi: 10.5527/wjn.v1.i3.69. PMID 24175244
- [Background] Saran R, Li Y, Robinson B, Ayanian J, Balkrishnan R, Bragg-Gresham J, Chen JT, Cope E, Gipson D, He K, Herman W, Heung M, Hirth RA, Jacobsen SS, Kalantar-Zadeh K, Kovesdy CP, Leichtman AB, Lu Y, Molnar MZ, Morgenstern H, Nallamothu B, O'Hare AM, Pisoni R, Plattner B, Port FK, Rao P, Rhee CM, Schaubel DE, Selewski DT, Shahinian V, Sim JJ, Song P, Streja E, Kurella Tamura M, Tentori F, Eggers PW, Agodoa LY, Abbott KC. US Renal Data System 2014 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2015 Jul;66(1 Suppl 1):Svii, S1-305. doi: 10.1053/j.ajkd.2015.05.001. No abstract available. PMID 26111994
- [Background] Office NRoD: Trends in Chronic Kidney Failure Stage 5 in Singapore 2012 / 2013. In.
- [Background] Rajan DK, Bunston S, Misra S, Pinto R, Lok CE. Dysfunctional autogenous hemodialysis fistulas: outcomes after angioplasty--are there clinical predictors of patency? Radiology. 2004 Aug;232(2):508-15. doi: 10.1148/radiol.2322030714. PMID 15286321
- [Background] Manninen HI, Kaukanen ET, Ikaheimo R, Karhapaa P, Lahtinen T, Matsi P, Lampainen E. Brachial arterial access: endovascular treatment of failing Brescia-Cimino hemodialysis fistulas--initial success and long-term results. Radiology. 2001 Mar;218(3):711-8. doi: 10.1148/radiology.218.3.r01mr38711. PMID 11230644
- [Background] Heye S, Maleux G, Vaninbroukx J, Claes K, Kuypers D, Oyen R. Factors influencing technical success and outcome of percutaneous balloon angioplasty in de novo native hemodialysis arteriovenous fistulas. Eur J Radiol. 2012 Sep;81(9):2298-303. doi: 10.1016/j.ejrad.2011.09.004. Epub 2011 Sep 28. PMID 21955605
- [Background] Haskal ZJ, Trerotola S, Dolmatch B, Schuman E, Altman S, Mietling S, Berman S, McLennan G, Trimmer C, Ross J, Vesely T. Stent graft versus balloon angioplasty for failing dialysis-access grafts. N Engl J Med. 2010 Feb 11;362(6):494-503. doi: 10.1056/NEJMoa0902045. PMID 20147715
- [Background] Shemesh D, Goldin I, Zaghal I, Berlowitz D, Raveh D, Olsha O. Angioplasty with stent graft versus bare stent for recurrent cephalic arch stenosis in autogenous arteriovenous access for hemodialysis: a prospective randomized clinical trial. J Vasc Surg. 2008 Dec;48(6):1524-31, 1531.e1-2. doi: 10.1016/j.jvs.2008.07.071. Epub 2008 Oct 1. PMID 18829240
- [Background] Salman L, Asif A. Stent graft for nephrologists: concerns and consensus. Clin J Am Soc Nephrol. 2010 Jul;5(7):1347-52. doi: 10.2215/CJN.02380310. Epub 2010 May 27. PMID 20507955
- [Background] Allon M. Current management of vascular access. Clin J Am Soc Nephrol. 2007 Jul;2(4):786-800. doi: 10.2215/CJN.00860207. Epub 2007 May 30. PMID 17699495
- [Background] Katsanos K, Karnabatidis D, Kitrou P, Spiliopoulos S, Christeas N, Siablis D. Paclitaxel-coated balloon angioplasty vs. plain balloon dilation for the treatment of failing dialysis access: 6-month interim results from a prospective randomized controlled trial. J Endovasc Ther. 2012 Apr;19(2):263-72. doi: 10.1583/11-3690.1. PMID 22545894
- [Background] Kennedy SA, Mafeld S, Baerlocher MO, Jaberi A, Rajan DK. Drug-Coated Balloon Angioplasty in Hemodialysis Circuits: A Systematic Review and Meta-Analysis. J Vasc Interv Radiol. 2019 Apr;30(4):483-494.e1. doi: 10.1016/j.jvir.2019.01.012. Epub 2019 Mar 8. PMID 30857987
- [Background] Katsanos K, Spiliopoulos S, Kitrou P, Krokidis M, Karnabatidis D. Risk of Death Following Application of Paclitaxel-Coated Balloons and Stents in the Femoropopliteal Artery of the Leg: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Am Heart Assoc. 2018 Dec 18;7(24):e011245. doi: 10.1161/JAHA.118.011245. PMID 30561254
- [Background] Updated CIRSE Position Statement on the use of paclitaxel-coated balloons and stents in peripheral arterial disease.https://www.cirse.org/research/current-updates/
- [Background] UPDATE: Treatment of Peripheral Arterial Disease with Paclitaxel-Coated Balloons and Paclitaxel-Eluting Stents Potentially Associated with Increased Mortality - Letter to Health Care Providers. https://www.fda.gov/medical-devices/letters-health-care-providers/update-treatment-peripheral-arterial-disease-paclitaxel-coated-balloons-and-paclitaxel-eluting
- [Background] Clever YP, Peters D, Calisse J, Bettink S, Berg MC, Sperling C, Stoever M, Cremers B, Kelsch B, Bohm M, Speck U, Scheller B. Novel Sirolimus-Coated Balloon Catheter: In Vivo Evaluation in a Porcine Coronary Model. Circ Cardiovasc Interv. 2016 Apr;9(4):e003543. doi: 10.1161/CIRCINTERVENTIONS.115.003543. PMID 27069105
- [Background] Verheye S, Vrolix M, Kumsars I, Erglis A, Sondore D, Agostoni P, Cornelis K, Janssens L, Maeng M, Slagboom T, Amoroso G, Jensen LO, Granada JF, Stella P. The SABRE Trial (Sirolimus Angioplasty Balloon for Coronary In-Stent Restenosis): Angiographic Results and 1-Year Clinical Outcomes. JACC Cardiovasc Interv. 2017 Oct 23;10(20):2029-2037. doi: 10.1016/j.jcin.2017.06.021. Epub 2017 Sep 27. PMID 28964764
- [Derived] Pang SC, Tan RY, Choke E, Ho J, Tay KH, Gogna A, Irani FG, Zhuang KD, Toh L, Chan S, Krishnan P, Lee KA, Leong S, Lo R, Patel A, Tan BS, Too CW, Chua J, Tng RKA, Tang TY, Chng SP, Chong TT, Tay HT, Yap HY, Wong J, Dharmaraj RB, Ng JJ, Gopinathan A, Loh EK, Ong SJ, Yoong G, Tay JS, Chong KY, Tan CS. SIroliMus coated angioPlasty versus plain balloon angioplasty in the tREatment of dialySis acceSs dysfunctION (IMPRESSION): study protocol for a randomized controlled trial. Trials. 2021 Dec 20;22(1):945. doi: 10.1186/s13063-021-05920-3. PMID 34930401